CLINICAL TRIAL: NCT05684952
Title: The Efficacy and Safety of a Chinese Herbal Medicine (Shenlingcao Oral Liquid) for Treating Long COVID Associated Fatigue：a Double-blinded, Placebo-controlled, Randomized Clinical Trial
Brief Title: The Efficacy and Safety of a Chinese Herbal Medicine for Long COVID Associated Fatigue
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Jiangzhong Pharmaceutical Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, ZhaoXiang Bian, Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LongCov-fatigue CHM
Record Dates: First submitted 2023-01-11; First posted 2023-01-13 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Long COVID
Keywords: fatigue; Chinese herbal medicine
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue

STUDY DESIGN:
Intervention Model Description: A double-blinded, placebo-controlled, randomized clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Subjects need to take the Chinese herbal medicine (Shenlingcao oral liquid) 200 ml twice per day for 4 weeks. Shenlingcao oral solution is comprised of American Ginseng (Panacis Quinquefolii Radix), Lucid Ganoderma (Ganoderma), Rose (Rosae Rugosae Flos) and fermented Cordyceps powder.
  Interventions: Drug: Shenlingcao Oral Liquid
- Control group (Placebo Comparator): Subjects need to take the placebo of Shenlingcao oral liquid 200 ml twice per day for 4 weeks.
  Interventions: Drug: Shenlingcao Oral Liquid

INTERVENTIONS:
Drug: Shenlingcao Oral Liquid — Shenlingcao oral liquid (200ml/bottle) is comprised of American Ginseng (Panacis Quinquefolii Radix), Lucid Ganoderma (Ganoderma), Rose (Rosae Rugosae Flos) and fermented Cordyceps powder.
  Other Names: placebo of Shenlingcao Oral Liquid

SUMMARY:
This is a randomized, double-blinded, placebo-controlled clinical trial to determine the efficacy and safety of a Chinese herbal medicine (Shenlingcao oral liquid) for treating long COVID associated fatigue.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled clinical trial to determine the efficacy and safety of a Chinese herbal medicine (Shenlingcao oral liquid) for treating long COVID associated fatigue. Our target population is adults (18-65 years old) with a COVID-19 infection history and have moderate to severe fatigue symptom at least 4 weeks after infection. The total sample size is 152. All participants will be randomly attributed to treatment group or placebo group in 1:1 ratio. The treatment duration is 4-week, and the follow-up period is also 4 weeks. Shenlingcao oral solution has been registered and marketed in mainland China, it is a safe product and pervious studies suggested it has anti-fatigue function. The primary efficacy outcome is the change of scores of Chalder fatigue scale (0-33 points) after 4-week treatment. The primary safety outcome is the number of adverse events. This study will be conducted in Hong Kong Baptist University Mr. & Mrs. Chan Hon Yin Chinese Medicine Specialty Clinic and Good Clinical Practice Centre.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years adults
2. Fulfill the long COVID diagnostic criteria by Centers for Disease Control and Prevention (CDC)
3. Chalder fatigue scale (0-11) not less than 4

Exclusion Criteria:

1. Have any medical history that may cause fatigue before COVID-19 infection, which include but not limited to cardiovascular diseases, chronic lung diseases, dyspnea, cognitive diseases, psychological diseases, chronic liver or renal diseases, cancer, etc.
2. Must chronically taking medicines that may affect the study results.
3. Severe obesity (BMI not less than 45)
4. Alcoholism or drug abuse
5. Allergy to Chinese medicine
6. Pregnancy, or plan to be pregnant, or lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue: Change of scores in Chalder fatigue scale (0-33 points) | 4 weeks
  The Chalder fatigue scale (CFQ) is a questionnaire to measure the severity of tiredness in fatiguing illnesses.

SECONDARY OUTCOMES:
Insomnia: Change of scores in Insomnia Severity Index (ISI) | 4 weeks
  The Insomnia Severity Index (ISI) is a brief instrument that was designed to assess the severity of both nighttime and daytime components of insomnia.
Quality of life: Change of scores in 36-Item Short Form Survey (SF-36) | 4 weeks
  The 36-Item Short Form Survey (SF-36) is an outcome measure instrument that is often used, well-researched, self-reported measure of health.
Mood: Change of scores in The Hospital Anxiety and Depression Scale (HADS) | 4 weeks
  HADS was found to perform well in assessing the symptom severity and caseness of anxiety disorders and depression
Muscle strength: Change of Hand Grip Strength (HGS) | 4 weeks
  Handgrip strength (HGS) is a simple and reliable measurement of maximum voluntary muscle strength. It is an important tool for diagnosing sarcopenia and is widely used as a single indicator to represent overall muscle strength
Long Covid related symptoms | 4 weeks
  Assessed by the self-reporting severity of 27 common symptoms after COVID-19 infection.
Safety: number of adverse events | 4 weeks
  Assessed by number of adverse events or side effects
Exploratory outcome: Immunology analysis | 4 weeks
  Assessed by the change of important immune index in serumImmune index
Exploratory outcome: Gut microbiota analysis | 4 weeks
  Assessed by the change of gut microbiota composition and its metabolimics.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Baptist University Chinese Medicine Clinic, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided